CLINICAL TRIAL: NCT03976427
Title: Changing How the Brain Responds When Making Decisions: Translating Neuroscience to Population Health
Brief Title: Translating Neuroscience to Population Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00142526
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a guided imagery exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided Imagery (Experimental): Participants will listen to a guided imagery recording
  Interventions: Behavioral: Guided Imagery

INTERVENTIONS:
Behavioral: Guided Imagery — The guided imagery exercise asks participants to think about positive associations with healthy foods and imagine their future healthy selves.

SUMMARY:
The current study will examine the relationship between brain responses and a guided imagery exercise in overweight and obese individuals. Results of this work are highly relevant to public health because they employ neuroimaging methods to understand food decision-making. Findings from this study will inform health decision making and holds great potential for future translation across multiple health behaviors and scalable interventions to impact population health

DETAILED DESCRIPTION:
Negative health behaviors (e.g. overeating, smoking) are associated with increased negative health outcomes. Engaging in healthy behaviors is not always rewarding (e.g. carrot vs. cake). Neural models of healthy behaviors focus on the balance between reward and regulation brain regions. The current pilot application examines the engagement of these regions during the evaluation of food and nonfood cues before and after a guided imagery exercise targeting positive associations with food and regulation.

The long-term goal is to understand the interaction between positive associations with healthy foods and thinking about future rewards may influence healthy decision-making. The objective of the current study is to empirically test the combined effects of positive affect and positive episodic future thinking on brain activation.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 25 to 55 kg/m2
* right-handed
* not currently dieting or attempting to lose weight.

Exclusion Criteria:

* serious medical illness unsuitable for the magnetic resonance imaging scanner based on best clinical judgment
* any neurologic or current psychiatric diagnosis
* currently taking anti-seizure medication
* history of concussion
* left-handedness
* risk for hazard due to magnetic fields such as metal in the body surgically or accidentally
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Brain Activation in Self-Regulation Brain Regions | 1 hour
  Functional Magnetic Resonance Imaging will measure brain activation changes in self-regulation brain regions including the dorsolateral prefrontal cortex, dorsomedial prefrontal cortex and anterior cingulate cortex when participants view healthy compared to unhealthy food images before and after the guided imagery exercise
Brain Activation in Reward Brain Regions | 1 hour
  Functional Magnetic Resonance Imaging will measure brain activation changes in reward brain regions including the ventromedial prefrontal cortex and striatum when participants view healthy compared to unhealthy food images before and after the guided imagery exercise

SECONDARY OUTCOMES:
Food Choice | 1 hour
  Observational preference for healthy compared to unhealthy food choices measured by the number of healthy and unhealthy foods selected following the guided imagery exercise
Food Demand | 1 hour
  Behavioral changes in demand for healthy compared to unhealthy foods will be measured by asking participants to indicate how healthy and unhealthy food items they would eat in a day if the items were freely available

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for primary outcomes will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 1-year after study completion
Access Criteria: Researchers may contact the Principal Investigator to request the data and will be required to sign research sharing agreements with the institution before gaining access.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT03976427/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03976427/ICF_001.pdf